CLINICAL TRIAL: NCT04074928
Title: A Phase 3, Randomized, Observer-Blind, Multicenter, Noninferiority Study to Evaluate Safety and Immunogenicity of a Cell-Based Quadrivalent Subunit Influenza Virus Vaccine (QIVc) and a United States Licensed Quadrivalent Influenza Virus Vaccine (QIV) in Healthy Subjects 6 Months Through 47 Months
Brief Title: Safety and Immunogenicity Study of QIVc in Healthy Pediatric Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V130_10; 2020-002785-13 (EudraCT Number)
Record Dates: First submitted 2019-08-27; First posted 2019-08-30 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Influenza; Human; Virus Diseases
Keywords: Influenza; RNA Virus; WHO Strains
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The trial is designed as an observer-blind study. During the treatment period of the study designated unblinded nurse(s), physician(s), or other qualified health care professional will be responsible for administering the study vaccine to the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QIVc (Experimental): Cell-derived Quadrivalent Influenza Vaccine containing 2 influenza type A strains and 2 influenza type B strains
  Interventions: Biological: QIVc
- Comparator QIV (Active Comparator): Comparator Quadrivalent Influenza Vaccine containing 2 influenza type A strains and 2 influenza type B strains
  Interventions: Biological: Comparator QIV

INTERVENTIONS:
Biological: QIVc — Previously vaccinated subjects received a 0.5 mL intramuscular dose of QIVc on Day 1; not previously vaccinated subjects received a 0.5 mL intramuscular dose of QIVc on Day 1 and Day 29.
  Other Names: Flucelvax Quadrivalent
  Arms: QIVc
Biological: Comparator QIV — Previously vaccinated subjects received a dose of Comparator QIV on Day 1; not previously vaccinated subjects received a dose of Comparator QIV on Day 1 and Day 29. Subjects 6 months through 35 months of age received a 0.25 mL intramuscular dose of Comparator QIV; subjects 36 months through 47 months of age received a 0.5 mL intramuscular dose of Comparator QIV.
  Other Names: Afluria Quadrivalent
  Arms: Comparator QIV

SUMMARY:
This phase 3 clinical study is a randomized, observer-blind, comparator-controlled, multicenter study of QIVc versus a US-licensed comparator QIV in children 6 months through 47 months of age. The purpose of this study is to demonstrate that vaccination with QIVc elicits an immune response that is noninferior to that of a US-licensed comparator QIV containing the same virus strains, in children 6 months through 47 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of 6 through 47 months of age on the day of informed consent.
* Individuals whose parent(s)/Legally Acceptable Representative (LAR) have voluntarily given written informed consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
* Individuals who can comply with study procedures including follow-up
* Individual is in generally good health as per the Investigator's medical judgement

Exclusion Criteria:

* Acute (severe) febrile illness
* History of any anaphylaxis, serious vaccine reactions or hypersensitivity, including allergic reactions, to any component of vaccine or medical equipment whose use is foreseen in this study
* A known history of Guillain-Barre Syndrome or other demyelinating diseases such as encephalomyelitis and transverse myelitis
* Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study
* Received influenza vaccination or has had documented influenza disease in the last 6 months prior to informed consent.

Ages: 6 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2414 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Seqirus
Locations (47):
- United States (47):
  - 84035 CCR Research, Mobile, Alabama
  - 84040 Southland Clnical Research Center, Anaheim, California
  - 84044 Premier Health Research Center, Downey, California
  - 84028 Orange County Research Institute, Ontario, California
  - 84029 Center for Clinical Trials, Paramount, California
  - 84012 Benchmark Research, Sacramento, California
  - 84006 California Research Foundation, San Diego, California
  - 84001 Acevedo Clincal Research Associates, Miami, Florida
  - 84005 Sunshine Research Center, Opa-locka, Florida
  - 84052 Tekton Research, Chamblee, Georgia
  - 84036 Advanced Clinical Research, Meridian, Idaho
  - 84027 Heartland Research Associates, El Dorado, Kansas
  - 84020 Heartland Research Associates, Newton, Kansas
  - 84014 Heartland Research Associates, Wichita, Kansas
  - 84026 Heartland Research Associates, Wichita, Kansas
  - 84041 Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - 84009 Bluegrass Clinical Research Inc., Louisville, Kentucky
  - 84008 Meridian Clinical Research, Baton Rouge, Louisiana
  - 84046 ACC Pediatric Research, Haughton, Louisiana
  - 84004 Benchmark Research, Metairie, Louisiana
  - 84022 Med Pharmics, Metairie, Louisiana
  - 84053 MedPharmics, Gulfport, Mississippi
  - 84051 Office of Craig A. Spiegel, Bridgeton, Missouri
  - 84016 Center for Pharmaceutical Research, Kansas City, Missouri
  - 84037 Meridian Clinical Research, Norfolk, Nebraska
  - 84017 Meridian Clinical Research, Omaha, Nebraska
  - 84033 Med Pharmics, Albuquerque, New Mexico
  - 84013 Regional Clinical Research, Binghamton, New York
  - 84045 Dayton Clinical, Dayton, Ohio
  - 84003 PriMed Clinical Research, Dayton, Ohio
  - 84015 Meridian Clinical Research, Dakota Dunes, South Dakota
  - 84032 Clinical Research Associates, Nashville, Tennessee
  - 84007 Benchmark Research, Austin, Texas
  - 84023 Ventavia Research Group, Fort Worth, Texas
  - 84042 Universtiy of North Texas Health Science Center, Fort Worth, Texas
  - 84043 Benchmark Research, Fort Worth, Texas
  - 84047 Ventavia Research Group, Houston, Texas
  - 84011 West Houston Clinical Research, Houston, Texas
  - 84019 Ventavia Research Group, Keller, Texas
  - 84021 Benchmark Research, San Angelo, Texas
  - 84002 Tekton Research, San Antonio, Texas
  - 84025 Pediatric Healthcare of NW Houston, Tomball, Texas
  - 84018 Tanner Clinic, Layton, Utah
  - 84050 JBR Clinical Research Group, Salt Lake City, Utah
  - 84048 J. Lewis Research/Foothill Family Clinic South, Salt Lake City, Utah
  - 84031 Advanced Clinical Research, West Jordan, Utah
  - 84039 Pediatric Research of Charlottesville, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Essink BJ, Heeringa M, Jeanfreau RJ, Finn D, Matassa V, Edelman J, Hohenboken M, Molrine D. Safety and Immunogenicity of Cell-Based Quadrivalent Influenza Vaccine: A Randomized Trial. Pediatrics. 2022 Nov 1;150(5):e2022057509. doi: 10.1542/peds.2022-057509. PMID 36214072

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in the 2019/2020 Northern Hemisphere influenza season from 47 centers in the United States.
Pre-assignment Details: In total, 2414 subjects were enrolled in the study.
Period: Overall Study
Arm/Group | QIVc | Comparator QIV
Started | 1605 | 809
Received Study Vaccine | 1597 | 805
Completed | 1370 | 710
Not Completed | 235 | 99

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS), defined as all enrolled subjects who were randomized and received a study vaccination.
Groups:
- Total: Total of all reporting groups
Arm/Group | QIVc | Comparator QIV | Total
Number analyzed (Participants) | 1597 | 805 | 2402
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1597 | 805 | 2402
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 28.1 (11.54) | 28.2 (11.63) | 28.1 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 794 | 399 | 1193
  Male | 803 | 406 | 1209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 434 | 226 | 660
  Not Hispanic or Latino | 1160 | 575 | 1735
  Unknown or Not Reported | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 11 | 22
  Asian | 13 | 8 | 21
  Native Hawaiian or Other Pacific Islander | 8 | 6 | 14
  Black or African American | 455 | 209 | 664
  White | 1039 | 539 | 1578
  Other | 71 | 32 | 103
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1597 | 805 | 2402

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity Endpoint: Geometric Mean Titer (GMT) and GMT Ratio Against the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by Hemagglutination Inhibition (HAI) Assay Using Cell-derived Target Viruses
Description: The GMT ratio is defined as the geometric mean of the postvaccination (28 days after last vaccination) HAI titer for the Comparator QIV divided by the geometric mean of the postvaccination HAI titer for QIVc.
Time Frame: Day 29 for previously vaccinated subjects; Day 57 for not previously vaccinated subjects
Population: Per Protocol Set (PPS): All subjects in the FAS who received vaccine on Day 1, provided serology specimens which yielded valid serology assay results from both Day 1 and Day 29 (previously vaccinated subjects) or Day 1 and Day 57 (not previously vaccinated subjects) and for whom there was no protocol deviation that was medically assessed as having potential to impact the immunogenicity results.
  1092 and 575 subjects in the QIVc and Comparator QIV groups had HAI assay data for this outcome.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | QIVc | Comparator QIV
Number analyzed (Participants) | 1092 | 575
Titer
  A/H1N1 | 78.0 [70.75 to 86.03] | 57.3 [50.76 to 64.63]
  B/Yamagata | 35.6 [32.93 to 38.58] | 26.0 [23.54 to 28.63]
  B/Victoria | 22.4 [20.70 to 24.19] | 19.6 [17.81 to 21.58]
Statistical Analysis 1: Comparison: QIVc vs Comparator QIV; Non-inferiority, A/H1N1, GMT ratio, Day 29/57 Non-inferiority of the Day 29/57 immune response to the A/H1N1 vaccine strain calculated by GMT ratio (Comparator QIV GMT divided by QIVc GMT); Test type: Non-Inferiority — The non-inferiority criterion was that the upper limit of the 2-sided 95% CI did not exceed the prespecified non-inferiority margin of 1.5 for the Day 29/57 GMT ratio (adjusted analysis); GMT ratio = 0.73, 95% CI 2-sided [0.645 to 0.836]
Statistical Analysis 2: Comparison: QIVc vs Comparator QIV; Non-inferiority, B/Yamagata, GMT ratio, Day 29/57 Non-inferiority of the Day 29/57 immune response to the B/Yamagata vaccine strain calculated by GMT ratio (Comparator QIV GMT divided by QIVc GMT); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMT ratio = 0.73, 95% CI 2-sided [0.656 to 0.809]
Statistical Analysis 3: Comparison: QIVc vs Comparator QIV; Non-inferiority, B/Victoria, GMT ratio, Day 29/57 Non-inferiority of the Day 29/57 immune response to the B/Victoria vaccine strain calculated by GMT ratio (Comparator QIV GMT divided by QIVc GMT); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMT ratio = 0.88, 95% CI 2-sided [0.791 to 0.972]

2. Primary Outcome: Immunogenicity Endpoint: Seroconversion Rates (SCR) and Differences in SCR Against the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by HAI Assay Using Cell-derived Target Viruses
Description: The SCR is defined as the percentage of subjects with either a prevaccination HAI titer <1:10 and a postvaccination HAI titer ≥1:40, or a prevaccination HAI titer ≥1:10 and a ≥4-fold increase in postvaccination HAI titer.
  The SCR difference is defined as the Comparator QIV SCR minus the QIVc SCR.
Time Frame: Day 1 to Day 29 for previously vaccinated subjects; Day 1 to Day 57 for not previously vaccinated subjects
Population: PPS (1092 and 575 subjects in the QIVc and Comparator QIV groups, respectively, had HAI assay data for this outcome)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | QIVc | Comparator QIV
Number analyzed (Participants) | 1092 | 575
Percentage of participants
  A/H1N1 | 58.24 [55.25 to 61.19] | 46.78 [42.64 to 50.96]
  B/Yamagata | 46.52 [43.53 to 49.53] | 31.65 [27.87 to 35.63]
  B/Victoria | 30.31 [27.60 to 33.13] | 24.35 [20.89 to 28.07]
Statistical Analysis 1: Comparison: QIVc vs Comparator QIV; Non-inferiority, A/H1N1, SCR difference, Day 29/57 Non-inferiority of the immune response to the A/H1N1 vaccine strain by SCR difference (Comparator QIV SCR minus QIVc SCR); Test type: Non-Inferiority — The non-inferiority criterion was that the upper limit of the 2-sided 95% CI did not exceed the prespecified non-inferiority margin of 10% for the Day 29/57 SCR difference; SCR difference = -11.46, 95% CI 2-sided [-16.447 to -6.423]
Statistical Analysis 2: Comparison: QIVc vs Comparator QIV; Non-inferiority, B/Yamagata, SCR difference, Day 29/57 Non-inferiority of the immune response to the B/Yamagata vaccine strain by SCR difference (Comparator QIV SCR minus QIVc SCR); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; SCR difference = -14.87, 95% CI 2-sided [-19.610 to -9.983]
Statistical Analysis 3: Comparison: QIVc vs Comparator QIV; Non-inferiority, B/Victoria, SCR difference, Day 29/57 Non-inferiority of the immune response to the B/Victoria vaccine strain by SCR difference (Comparator QIV SCR minus QIVc SCR); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; SCR difference = -5.96, 95% CI 2-sided [-10.327 to -1.440]

3. Primary Outcome: Immunogenicity Endpoint: GMT and GMT Ratio Against the A/H3N2 Vaccine Strain by Microneutralization (MN) Assay Using Cell-derived Target Viruses
Description: The GMT ratio is defined as the geometric mean of the postvaccination (28 days after last vaccination) MN titer for the Comparator QIV divided by the geometric mean of the postvaccination MN titer for QIVc.
Time Frame: Day 29 for previously vaccinated subjects; Day 57 for not previously vaccinated subjects
Population: PPS (1078 and 572 subjects in the QIVc and Comparator QIV groups, respectively, had MN assay data for this outcome)
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | QIVc | Comparator QIV
Number analyzed (Participants) | 1078 | 572
Titer | 23.1 [21.21 to 25.12] | 23.9 [21.57 to 26.57]
Statistical Analysis 1: Comparison: QIVc vs Comparator QIV; Non-inferiority, A/H3N2, GMT ratio, Day 29/57 Non-inferiority of the Day 29/57 immune response to the A/H3N2 vaccine strain calculated by GMT ratio (Comparator QIV GMT divided by QIVc GMT); Test type: Non-Inferiority — The noninferiority criterion was that the upper limit of the 2-sided 95% CI did not exceed the prespecified noninferiority margin of 1.5 for the Day 29/57 GMT ratio (adjusted analysis); GMT ratio = 1.04, 95% CI 2-sided [0.927 to 1.160]

4. Primary Outcome: Immunogenicity Endpoint: SCR and Difference in SCR Against the A/H3N2 Vaccine Strain by MN Assay Using Cell-derived Target Viruses
Description: The SCR is defined as the percentage of subjects with either a prevaccination MN titer <1:10 and a postvaccination MN titer ≥1:40, or a prevaccination MN titer ≥1:10 and a ≥4-fold increase in postvaccination MN titer.
  The SCR difference is defined as the Comparator QIV SCR minus the QIVc SCR.
Time Frame: Day 1 to Day 29 for previously vaccinated subjects; Day 1 to Day 57 for not previously vaccinated subjects
Population: PPS (1078 and 572 subjects in the QIVc and Comparator QIV groups, respectively, had MN assay data for this outcome)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | QIVc | Comparator QIV
Number analyzed (Participants) | 1078 | 572
Percentage of participants | 27.64 [24.99 to 30.42] | 30.77 [27.01 to 34.73]
Statistical Analysis 1: Comparison: QIVc vs Comparator QIV; Non-inferiority, A/H3N2, SCR difference, Day 29/57 Non-inferiority of the immune response to the A/H3N2 vaccine strain by SCR difference (Comparator QIV SCR minus QIVc SCR); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; SCR difference = 3.13, 95% CI 2-sided [-1.443 to 7.812]

5. Secondary Outcome: Immunogenicity Endpoint: GMT and GMT Ratio Against the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by HAI Assay Using Egg-derived Target Viruses
Description: as for outcome 1
Time Frame: Day 1 and Day 29 for previously vaccinated subjects; Day 1 and Day 57 for not previously vaccinated subjects
Population: PPS (1092 and 575 subjects in the QIVc and Comparator QIV groups, respectively, had HAI assay data for this outcome)
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | QIVc | Comparator QIV
Number analyzed (Participants) | 1092 | 575
Titer
  A/H1N1 Day 1 HAI GMT | 14.0 [12.54 to 15.74] | 13.9 [12.11 to 16.04]
  A/H1N1 Day 29/57 HAI GMT | 92.2 [83.62 to 101.71] | 82.9 [73.51 to 93.58]
  B/Yamagata Day 1 HAI GMT | 6.7 [6.33 to 7.16] | 6.7 [6.23 to 7.26]
  B/Yamagata Day 29/57 HAI GMT | 23.0 [21.21 to 24.89] | 24.7 [22.39 to 27.26]
  B/Victoria Day 1 HAI GMT | 6.1 [5.77 to 6.38] | 6.0 [5.68 to 6.43]
  B/Victoria Day 29/57 HAI GMT | 13.6 [12.58 to 14.61] | 14.8 [13.46 to 16.19]
Statistical Analysis 1: Comparison: QIVc vs Comparator QIV; A/H1N1, GMT ratio, Day 29/57; Test type: Other — No formal statistical testing was planned for this secondary outcome measure; GMT ratio = 0.90, 95% CI 2-sided [0.790 to 1.024]
Statistical Analysis 2: Comparison: QIVc vs Comparator QIV; B/Yamagata, GMT ratio, Day 29/57; Test type: Other — No formal statistical testing was planned for this secondary outcome measure; GMT ratio = 1.08, 95% CI 2-sided [0.968 to 1.195]
Statistical Analysis 3: Comparison: QIVc vs Comparator QIV; B/Victoria, GMT ratio, Day 29/57; Test type: Other — No formal statistical testing was planned for this secondary outcome measure; GMT ratio = 1.09, 95% CI 2-sided [0.986 to 1.202]

6. Secondary Outcome: Immunogenicity Endpoint: SCR and Difference in SCR Against the A/H1N1, B/Victoria and B/ Yamagata Vaccine Strains by HAI Assay Using Egg-derived Target Viruses
Description: as for outcome 2
Time Frame: Day 1 to Day 29 for previously vaccinated subjects; Day 1 to Day 57 for not previously vaccinated subjects
Population: PPS (1092 and 575 subjects in the QIVc and Comparator QIV groups, respectively, had HAI assay data for this outcome)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | QIVc | Comparator QIV
Number analyzed (Participants) | 1092 | 575
Percentage of participants
  A/H1N1 HAI SCR | 58.52 [55.53 to 61.46] | 56.00 [51.83 to 60.10]
  B/Yamagata HAI SCR | 38.64 [35.74 to 41.61] | 38.61 [34.61 to 42.73]
  B/Victoria HAI SCR | 19.69 [17.37 to 22.17] | 20.87 [17.62 to 24.42]
Statistical Analysis 1: Comparison: QIVc vs Comparator QIV; A/H1N1, SCR difference, Day 29/57; Test type: Other — No formal statistical testing was planned for this secondary outcome measure; SCR difference = -2.52, 95% CI 2-sided [-7.526 to 2.461]
Statistical Analysis 2: Comparison: QIVc vs Comparator QIV; B/Yamagata, SCR difference, Day 29/57; Test type: Other — No formal statistical testing was planned for this secondary outcome measure; SCR difference = -0.04, 95% CI 2-sided [-4.912 to 4.911]
Statistical Analysis 3: Comparison: QIVc vs Comparator QIV; B/Victoria, SCR difference, Day 29/57; Test type: Other — No formal statistical testing was planned for this secondary outcome measure; SCR difference = 1.18, 95% CI 2-sided [-2.805 to 5.353]

7. Secondary Outcome: Immunogenicity Endpoint: GMT and GMT Ratio Against the A/H3N2 Vaccine Strain by MN Assay Using Egg-derived Target Viruses
Description: as for outcome 3
Time Frame: Day 1 and Day 29 for previously vaccinated subjects; Day 1 and Day 57 for not previously vaccinated subjects
Population: PPS (1079 and 572 subjects in the QIVc and Comparator QIV groups, respectively, had MN assay data for this outcome)
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | QIVc | Comparator QIV
Number analyzed (Participants) | 1079 | 572
Titer
  A/H3N2 Day 1 MN GMT | 12.9 [11.87 to 13.96] | 12.6 [11.42 to 13.95]
  A/H3N2 Day 29/57 MN GMT | 43.4 [39.58 to 47.52] | 44.7 [39.98 to 50.08]
Statistical Analysis 1: Comparison: QIVc vs Comparator QIV; A/H3N2, GMT ratio, Day 29/57; Test type: Other — No formal statistical testing was planned for this secondary outcome measure; GMT ratio = 1.03, 95% CI 2-sided [0.914 to 1.165]

8. Secondary Outcome: Immunogenicity Endpoint: SCR and Difference in SCR Against the A/H3N2 Vaccine Strain by MN Assay Using Egg-derived Target Viruses
Description: as for outcome 4
Time Frame: Day 1 to Day 29 for previously vaccinated subjects; Day 1 to Day 57 for not previously vaccinated subjects
Population: PPS (1079 and 572 subjects in the QIVc and Comparator QIV groups, respectively, had MN assay data for this outcome)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | QIVc | Comparator QIV
Number analyzed (Participants) | 1079 | 572
Percentage of participants | 37.44 [34.55 to 40.41] | 39.34 [35.31 to 43.47]
Statistical Analysis 1: Comparison: QIVc vs Comparator QIV; A/H3N2, SCR difference, Day 29/57; Test type: Other — No formal statistical testing was planned for this secondary outcome measure; SCR difference = 1.89, 95% CI 2-sided [-3.006 to 6.856]

9. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Ratio (GMR) Against the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by HAI Assay Using Cell-derived and Egg-derived Target Viruses
Description: GMR is defined as the geometric mean of the (within-subject) fold increase in serum HAI GMT postvaccination (Day 29/57) compared to prevaccination (Day 1).
Time Frame: Day 1 to Day 29 for previously vaccinated subjects; Day 1 to Day 57 for not previously vaccinated subjects
Population: PPS (1092 and 575 subjects in the QIVc and Comparator QIV groups, respectively, had HAI assay data for this outcome)
Measure: Number (95% Confidence Interval); unit: Geometric mean ratio
Arm/Group | QIVc | Comparator QIV
Number analyzed (Participants) | 1092 | 575
Geometric mean ratio
  A/H1N1 (cell) HAI GMR | 5.34 [4.834 to 5.910] | 3.97 [3.506 to 4.493]
  B/Yamagata (cell) HAI GMR | 4.12 [3.792 to 4.467] | 3.03 [2.735 to 3.348]
  B/Victoria (cell) HAI GMR | 2.65 [2.450 to 2.864] | 2.31 [2.100 to 2.548]
  A/H1N1 (egg) HAI GMR | 5.67 [5.117 to 6.290] | 5.11 [4.503 to 5.809]
  B/Yamagata (egg) HAI GMR | 3.04 [2.808 to 3.298] | 3.27 [2.964 to 3.615]
  B/Victoria (egg) HAI GMR | 2.14 [1.987 to 2.308] | 2.33 [2.126 to 2.558]

10. Secondary Outcome: Immunogenicity Endpoint: GMR Against the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by MN Assay Using Cell-derived and Egg-derived Target Viruses
Description: GMR is defined as the geometric mean of the (within-subject) fold increase in serum MN GMT postvaccination (Day 29/57) compared to prevaccination (Day 1).
Time Frame: Day 1 to Day 29 for previously vaccinated subjects; Day 1 to Day 57 for not previously vaccinated subjects
Population: PPS (A randomly selected subset of subjects; 195 and 122 subjects in the QIVc and Comparator QIV groups, respectively, had MN assay data for this outcome) The MN assays for A/H1N1, B/Yamagata, and B/Victoria strains were only evaluated for cell-derived target viruses. Data were not collected for egg-derived target viruses.
Measure: Number (95% Confidence Interval); unit: Geometric mean ratio
Arm/Group | QIVc | Comparator QIV
Number analyzed (Participants) | 195 | 122
Geometric mean ratio
  A/H1N1 (cell) MN GMR | 5.74 [4.356 to 7.573] | 4.29 [3.174 to 5.811]
  B/Yamagata (cell) MN GMR | 3.14 [2.561 to 3.854] | 2.86 [2.284 to 3.572]
  B/Victoria (cell) MN GMR | 1.88 [1.583 to 2.241] | 1.63 [1.344 to 1.966]
  A/H1N1 (egg) MN GMR: number analyzed (Participants) | 0 | 0
  B/Yamagata (egg) MN GMR: number analyzed (Participants) | 0 | 0
  B/Victoria (egg) MN GMR: number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Immunogenicity Endpoint: GMR Against the A/H3N2 Vaccine Strain by MN Assay Using Cell-derived and Egg-derived Target Viruses
Description: as for outcome 10
Time Frame: Day 1 to Day 29 for previously vaccinated subjects; Day 1 to Day 57 for not previously vaccinated subjects
Population: PPS (1078 and 572 subjects in the QIVc and Comparator QIV groups, respectively, had MN assay data for the outcome of GMR against the A/H3N2 vaccine strain by MN assay using cell-derived target viruses; 1079 and 572 subjects in the QIVc and Comparator QIV groups, respectively, had data for the outcome of GMR against the A/H3N2 vaccine strain by MN assay using egg-derived target viruses)
Measure: Number (95% Confidence Interval); unit: Geometric mean ratio
Arm/Group | QIVc | Comparator QIV
Number analyzed (Participants) | 1079 | 572
Geometric mean ratio
  A/H3N2 (cell) MN GMR: number analyzed (Participants) | 1078 | 572
  A/H3N2 (cell) MN GMR | 2.11 [1.940 to 2.298] | 2.19 [1.977 to 2.436]
  A/H3N2 (egg) MN GMR | 3.13 [2.856 to 3.431] | 3.22 [2.878 to 3.608]

12. Secondary Outcome: Safety Endpoint: Percentage of Subjects With Solicited Adverse Events (AEs)
Description: The percentage of subjects with at least one solicited AE Day 1 through Day 7 after any study vaccination.
Time Frame: Day 1 to Day 7 after each vaccination (Day 1 to Day 7 for previously vaccinated subjects; Day 1 to Day 7 and Day 29 to Day 35 for not previously vaccinated subjects)
Population: Solicited Safety Set, defined as all subjects in the FAS with any solicited AE data.
Measure: Count of Participants; unit: Participants
Arm/Group | QIVc | Comparator QIV
Number analyzed (Participants) | 1564 | 784
Participants
  Solicited AEs | 940 | 491
  Solicited Local AEs | 656 | 350
  Solicited Systemic AEs | 681 | 358
  Analgesic/Antipyretic Use | 240 | 136

13. Secondary Outcome: Safety Endpoint: Percentage of Subjects With Any Unsolicited AEs
Description: The percentage of subjects with at least one unsolicited AE from Day 1 to Day 29 for previously vaccinated subjects and from Day 1 to Day 57 for not previously vaccinated subjects.
  Related AEs = considered at least possibly related to study vaccination by the investigator; Severity = based on the greatest severity associated with a preferred term for a reported AE.
Time Frame: Day 1 to Day 29 for previously vaccinated subjects; Day 1 to Day 57 for not previously vaccinated subjects
Population: Unsolicited Safety Set, defined as all subjects in the FAS with any unsolicited AE data.
Measure: Count of Participants; unit: Participants
Arm/Group | QIVc | Comparator QIV
Number analyzed (Participants) | 1597 | 805
Participants
  Any AE | 418 | 207
  Any AE (Mild) | 308 | 164
  Any AE (Moderate) | 98 | 41
  Any AE (Severe) | 12 | 2
  Related AE | 70 | 36

14. Secondary Outcome: Safety Endpoint: Percentage of Subjects With Any Serious Adverse Events (SAEs), New Onset of Chronic Disease (NOCD) or AEs Leading to Withdrawal During the Entire Study Period
Description: The percentage of subjects with any SAE, NOCD or AE leading to withdrawal during the study period from Day 1 to Day 181 for previously vaccinated subjects or from Day 1 to Day 209 for not previously vaccinated subjects.
  Definitions:
  SAEs = AEs defined as any untoward medical occurrence that at any dose resulted in one or more of the following: 1. Death, 2. Life-threatening 3. Required/prolonged hospitalization 4. Persistent or significant disability/incapacity 5. congenital anomaly/or birth defect 6. An important and significant medical event that may not be immediately life threatening or resulting in death or hospitalization but, based on appropriate medical judgment, may jeopardize the subject or may require intervention to prevent one of the other outcomes listed above
Time Frame: Day 1 to Day 181 for previously vaccinated subjects; Day 1 to Day 209 for not previously vaccinated subjects
Population: Unsolicited Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | QIVc | Comparator QIV
Number analyzed (Participants) | 1597 | 805
Participants
  SAE | 15 | 7
  Related SAE | 0 | 0
  AE leading to study withdrawal | 3 | 0
  NOCD | 22 | 13
  Death | 2 | 0

ADVERSE EVENTS:
Time Frame: SAEs: Day 1 to Day 181 for previously vaccinated subjects; Day 1 to Day 209 for not previously vaccinated subjects Nonserious unsolicited AEs: Day 1 to Day 29 for previously vaccinated subjects; Day 1 to Day 57 for not previously vaccinated subjects Solicited AEs: Day 1 to Day 7 after each vaccination (Day 1 to Day 7 for previously vaccinated subjects; Day 1 to Day 7 and Day 29 to Day 35 for not previously vaccinated subjects)
Description: SAEs, nonserious unsolicited AEs, and solicited AEs are reported in this Adverse Events section.
Arm/Group | QIVc | Comparator QIV
All-Cause Mortality (participants affected / at risk) | 2/1597 | 0/805
Serious Adverse Events (participants affected / at risk) | 15/1597 | 7/805
Other Adverse Events (participants affected / at risk) | 926/1597 | 490/805
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QIVc (N=1597) | Comparator QIV (N=805)
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Seizure (Nervous system disorders) | 2 | 0
Unresponsive to stimuli (Nervous system disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Ligamentitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Bronchiolitis (Infections and infestations) | 1 | 3
Pneumonia (Infections and infestations) | 3 | 0
Rhinovirus infection (Infections and infestations) | 1 | 1
Abscess of eyelid (Infections and infestations) | 1 | 0
Adenoviral encephalitis (Infections and infestations) | 1 | 0
Enterovirus infection (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | QIVc (N=1597) | Comparator QIV (N=805)
Upper respiratory tract infection (Infections and infestations) | 59 | 44
Injection site induration (General disorders) | 270/1564 | 125/784
Injection site erythema (General disorders) | 403/1564 | 193/784
Injection site ecchymosis (General disorders) | 168/1564 | 85/784
Injection site tenderness (General disorders) | 436/1564 | 235/784
Change of eating habits (Metabolism and nutrition disorders) | 272/1564 | 138/784
Sleepiness (Nervous system disorders) | 420/1564 | 200/784
Vomiting/throwing up (Gastrointestinal disorders) | 106/1564 | 49/784
Diarrhea/loose stools (Gastrointestinal disorders) | 280/1564 | 128/784
Irritability (Psychiatric disorders) | 436/1564 | 232/784
Fever (≥38.0°C) (General disorders) | 107/1564 | 54/784

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT04074928/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT04074928/SAP_001.pdf